CLINICAL TRIAL: NCT03901274
Title: Patient Centered Enhancements in School Behavioral Health: A Randomized Trial
Brief Title: Patient Centered Enhancements in School Behavioral Health
Acronym: PSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Maryland, Baltimore (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Mark Weist, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00085951
Record Dates: First submitted 2019-03-29; First posted 2019-04-03 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Mental Health
Keywords: School-based services; Stakeholder Engagement; Middle School
MeSH Terms: conditions — Psychological Well-Being | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wellness Condition (Active Comparator): Participants in this condition will receive school-based behavioral health services from clinicians who are trained in the evidence-based Wellness Framework.
  Interventions: Behavioral: Wellness
- Partnership (Experimental): Participants in this condition will receive school-based behavioral health services from clinicians who are trained in the evidence-based Wellness framework. The clinicians in this condition will receive additional training on patient-centered enhancements called the Partnership intervention.
  Interventions: Behavioral: Partnership

INTERVENTIONS:
Behavioral: Wellness — The Wellness framework packages together evidence-based practices of family engagement, modular evidence-based practice, quality assurance, and implementation support. Depending on their time of enrollment, participants can be involved in this condition for one to three years. They will be asked to complete assessments during their therapy sessions periodically throughout the trial.
  Arms: Wellness Condition
Behavioral: Partnership — The two patient-centered enhancements are: enhancing mental health literacy and stigma reduction, and improving family-school-mental health partnerships. Depending on their time of enrollment, participants can be involved in this condition for one to three years. They will be asked to complete assessments during their therapy sessions periodically throughout the trial.
  Arms: Partnership

SUMMARY:
This study will evaluate whether the evidence-based Wellness framework paired with an evidence-based Partnership compared to Wellness alone will improve middle school students' social, emotional/behavioral, and academic functioning.

DETAILED DESCRIPTION:
The mental health needs of children and youth are well-documented as an under-addressed and significant public health need in the United States. A number of barriers prevent children, youth, and families from accessing behavioral health services in standard clinic settings, including lack of sufficient transportation, cost, and stigma related to receiving services. School behavioral health (SBH) programs-in which community mental health providers join school teams to better address the social, emotional/behavioral, and academic needs of students-are growing in the United States because of their ability to reach youth who need, but may not otherwise receive, services. However, these efforts are limited by a lack of patient and stakeholder engagement. This has commonly resulted in SBH programs not being implemented, implemented inconsistently, or underutilized. The study will compare an evidence-based Patient-Centered Enhancements (i.e., Partnership) intervention added to an evidence-based framework termed Wellness in a three-year intervention for students in middle schools. Investigators predict the addition of the Partnership intervention will improve school climate and enhance SBH services, resulting in significantly improved social, emotional/behavioral, and academic outcomes in students. The study has three aims:

1. Investigators will evaluate the extent to which Partnership increases the number of students and families receiving school behavioral health services and expressing satisfaction with services received.
2. Investigators will evaluate the impact of Partnership on students' social, emotional/behavioral, and academic outcomes throughout the course of the intervention period (sixth through eighth grade).

ELIGIBILITY:
Inclusion Criteria:

* Middle school student
* Receives school-based behavioral health services
* Parent of a middle school student
* Parent of a student receiving school-based behavioral health services
* Enrolled in a participating school

Exclusion Criteria:

* Not a middle school student
* Not receiving school-based behavioral health services
* Not a parent of a middle school student
* Does not have a child receiving school-based behavioral health services
* Not enrolled in a participating school

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2558 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Weist, Ph.D., Principal Investigator — University of South Carolina
Locations (3):
- United States (3):
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Medical University of South Carolina, Charleston, South Carolina
  - University of South Carolina, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Connors, E.H., Stephan, S.H., Lever, N., Ereshefsky, S., Mosby, A., & Bohnenkamp, J. (2016). A national initiative to advance school mental health performance measurement in the US. Advances in School Mental Health Promotion, 9(1), 50-69.
- [Background] Weist, M.D., Sander, M.A., Walrath, C., Link, B., Nabors, L., Adelsheim, S., ... & Carrillo, K. (2005). Developing principles for best practice in expanded school mental health. Journal of Youth and Adolescence, 34(1), 7-13.
- [Background] Kutcher S, Wei Y, Morgan C. Successful Application of a Canadian Mental Health Curriculum Resource by Usual Classroom Teachers in Significantly and Sustainably Improving Student Mental Health Literacy. Can J Psychiatry. 2015 Dec;60(12):580-6. doi: 10.1177/070674371506001209. PMID 26720827
- [Background] Mcluckie A, Kutcher S, Wei Y, Weaver C. Sustained improvements in students' mental health literacy with use of a mental health curriculum in Canadian schools. BMC Psychiatry. 2014 Dec 31;14:379. doi: 10.1186/s12888-014-0379-4. PMID 25551789
- [Background] Haine-Schlagel R, Roesch SC, Trask EV, Fawley-King K, Ganger WC, Aarons GA. The Parent Participation Engagement Measure (PPEM): Reliability and Validity in Child and Adolescent Community Mental Health Services. Adm Policy Ment Health. 2016 Sep;43(5):813-823. doi: 10.1007/s10488-015-0698-x. PMID 26520104
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Price CS, Spence SH, Sheffield J, Donovan C. The development and psychometric properties of a measure of social and adaptive functioning for children and adolescents. J Clin Child Adolesc Psychol. 2002 Mar;31(1):111-22. doi: 10.1207/S15374424JCCP3101_13. PMID 11845643
- [Background] Chorpita BF, Reise S, Weisz JR, Grubbs K, Becker KD, Krull JL; Research Network on Youth Mental Health. Evaluation of the Brief Problem Checklist: child and caregiver interviews to measure clinical progress. J Consult Clin Psychol. 2010 Aug;78(4):526-36. doi: 10.1037/a0019602. PMID 20658809
- [Background] Brener ND, Collins JL, Kann L, Warren CW, Williams BI. Reliability of the Youth Risk Behavior Survey Questionnaire. Am J Epidemiol. 1995 Mar 15;141(6):575-80. doi: 10.1093/oxfordjournals.aje.a117473. PMID 7900725
- [Background] Abrishami, G.F. & Warren, J.S. (2013). Therapeutic alliance and outcomes in children and adolescents served in a community mental health system. Journal of Child & Adolescent Behavior, 1(2), 1-7.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As defined here, students who enrolled in the project were engaged in clinical services with a school-based mental health therapist. For some outcome measures, we used schoolwide data (e.g., grades, discipline) for all students enrolled at participating schools. There, number of participants analyzed are much larger due to overall school enrollment.
Units Other Than Participants: Schools
Period: Overall Study
Arm/Group | Wellness Condition | Partnership
Started (Participants described here include students and one parent/caregiver who enrolled and remained in the study together. Students reported data independently of their caregiver.) | 1330; 10 Schools | 1228; 10 Schools
Completed | 1210; 10 Schools | 1098; 10 Schools
Not Completed | 120; 0 Schools | 130; 0 Schools
Not completed — Lost to Follow-up | 120 | 124
Not completed — Withdrawal by Subject | 0 | 6

BASELINE CHARACTERISTICS:
Population: Number includes students and one parent/caregiver per student. However, many caregivers did not complete the intake survey which asked for parent age; therefore the number of caregivers is lower than the number of students in each condition. This number represents individual students/caregivers who completed self-reported surveys, which were the data utilized for individual, student-level outcomes. School-level variables are represented by # of total students enrolled or # of schools.
Groups:
- Total: Total of all reporting groups
Arm/Group | Wellness Condition | Partnership | Total
Number analyzed (Participants) | 1330 | 1228 | 2558
Age, Categorical [Count of Participants; unit: Participants] — Population: Age analysis applies only to students, whose age was available for calculation. Parent/caregiver age is not available for analysis.
  Participants
    Students: number analyzed (Participants) | 665 | 614 | 1279
    Students: <=18 years | 665 | 614 | 1279
    Students: Between 18 and 65 years | 0 | 0 | 0
    Students: >=65 years | 0 | 0 | 0
    Parents/Caregivers: number analyzed (Participants) | 509 | 398 | 907
    Parents/Caregivers: <=18 years | 0 | 0 | 0
    Parents/Caregivers: Between 18 and 65 years | 489 | 382 | 871
    Parents/Caregivers: >=65 years | 20 | 16 | 36
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Student - Female | 323 | 291 | 614
  Student - Male | 280 | 270 | 550
  Student - Nonbinary / Gender Non-Conforming | 29 | 29 | 58
  Student - Missing or Prefer Not to Answer | 33 | 24 | 57
  Parent - Female | 471 | 392 | 863
  Parent - Male | 57 | 47 | 104
  Parent - Nonbinary / Gender Non-Conforming | 3 | 2 | 5
  Parent - Missing or Prefer Not to Answer | 134 | 173 | 307
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Each row represents a segment of the enrolled population: students or parent/caregiver. To report more accurately, we have separated these groups. It is important to note, to account for exceptionally high number of unknown/not reported ethnicity, this is due to an error in data collection. The survey did not distinguish between race and ethnicity, therefore respondents may have indicated a race (e.g., Black/African American) and no ethnicity. We assign these as ethnicity unknown.
  Participants
    Students: number analyzed (Participants) | 665 | 614 | 1279
    Students: Hispanic or Latino | 47 | 38 | 85
    Students: Not Hispanic or Latino | 0 | 0 | 0
    Students: Unknown or Not Reported | 618 | 576 | 1194
    Parent/Caregiver: number analyzed (Participants) | 665 | 614 | 1279
    Parent/Caregiver: Hispanic or Latino | 39 | 35 | 74
    Parent/Caregiver: Not Hispanic or Latino | 0 | 0 | 0
    Parent/Caregiver: Unknown or Not Reported | 626 | 579 | 1205
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: As above, we are reporting student demographics separately from parent, for increased clarity in describing the population that enrolled. Similarly, a respondent may have indicated Hispanic (which is an ethnicity but as collected, not separated from race as an option) and not selected any other identifier. Thus, these individuals are reported as having no reported race.
  Participants
    Students: number analyzed (Participants) | 665 | 614 | 1279
    Students: American Indian or Alaska Native | 2 | 3 | 5
    Students: Asian | 5 | 5 | 10
    Students: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Students: Black or African American | 313 | 248 | 561
    Students: White | 198 | 220 | 418
    Students: More than one race | 52 | 50 | 102
    Students: Unknown or Not Reported | 95 | 88 | 183
    Parents / Caregivers: number analyzed (Participants) | 665 | 614 | 1279
    Parents / Caregivers: American Indian or Alaska Native | 3 | 1 | 4
    Parents / Caregivers: Asian | 2 | 4 | 6
    Parents / Caregivers: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Parents / Caregivers: Black or African American | 266 | 186 | 452
    Parents / Caregivers: White | 198 | 182 | 380
    Parents / Caregivers: More than one race | 22 | 17 | 39
    Parents / Caregivers: Unknown or Not Reported | 173 | 224 | 397

OUTCOME MEASURES:

1. Primary Outcome: Change in Emotional/Behavioral Functioning of Students Receiving Services
Description: Brief Problem Checklist: 12-item questionnaire measuring externalizing and internalizing problems found in children age 7-13 years old. Responses are given using a 3-point Likert scale ranging from 0 (not true) to 2 (very true), with responses summed for a possible score ranging from 0 to 24. High scores indicate a worse outcome for respondents. Analysis included students who completed at least 80% of the items on the scale.
Time Frame: Baseline (intake) and at 3 months and 6 months post-intake
Population: Students and parents who responded to at least 80% of items on the measure at each timepoint were included for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wellness Condition | Partnership
Number analyzed (Participants) | 1146 | 982
score on a scale
  Intake-student: number analyzed (Participants) | 614 | 550
  Intake-student | 9.03 (4.82) | 9.21 (4.71)
  3 months post-student: number analyzed (Participants) | 452 | 387
  3 months post-student | 8.86 (4.80) | 8.94 (4.60)
  6 months post-student: number analyzed (Participants) | 385 | 327
  6 months post-student | 9.05 (4.93) | 8.36 (4.70)
  Intake-parent: number analyzed (Participants) | 532 | 432
  Intake-parent | 8.48 (5.02) | 8.97 (5.34)
  3 months post-parent: number analyzed (Participants) | 235 | 263
  3 months post-parent | 7.15 (4.74) | 8.42 (5.01)
  6 months post-parent: number analyzed (Participants) | 195 | 212
  6 months post-parent | 7.12 (4.68) | 7.63 (4.65)
Statistical Analysis 1: Comparison: Wellness Condition vs Partnership; Intent-to-treat on three month outcomes with intake (i.e. Pretest covariate); Test type: Superiority; Slope = -0.16, 95% CI 2-sided [-0.74 to 0.42], Standard Error of Mean 0.29 — Parameter estimated with full information maximum likelihood
Statistical Analysis 2: Comparison: Wellness Condition vs Partnership; Intent-to-treat on six month outcomes with intake (i.e. Pretest covariate); Test type: Superiority; Slope = -0.65, 95% CI 2-sided [-1.20 to -0.09], Standard Error of Mean 0.28 — Parameter estimated with full information maximum likelihood

2. Primary Outcome: Change in Discipline Rates
Description: Computed models for student referrals to in-school suspension (ISS). The primary estimate can be interpreted as the log count difference between the treatment and control, and the zero inflated parameter can be interpreted as the log odds of not belonging to the inflated zero latent class. The primary analysis answers the question "Did random assignment to the Partnership condition change the number of observed behaviors?" and the zero inflated parameter asks "Did random assignment to the Partnership condition change the odds of having any observed behaviors?".
Time Frame: Annually per academic year
Population: This number includes all students who were enrolled at each of the 20 participating schools, not only those who were engaged in clinical practice. Students did not actively consent into this analysis of administrative school record data. Only a small fraction of the schoolwide population enrolled in the study to provide self-reported data on behaviors and clinical outcomes; whereas this analysis was of whole-school data.
Measure: Number; unit: participants
Arm/Group | Wellness Condition | Partnership
Number analyzed (Participants) | 18653 | 18652
participants
  2019-2020 school year | 4646 | 4646
  2020-2021 school year | 4555 | 4554
  2021-2022 school year | 4633 | 4633
  2022-2023 school year | 4819 | 4819

3. Primary Outcome: Change in Perceptions of School Climate
Description: School Climate Survey (SCS): a free, online climate survey from the US Department of Education (ED). The SCS is a 73-item questionnaire for students and an 83-item questionnaire for school instructional and non-instructional staff on a 4 point scale ranging from 1 "Strongly Agree" to 4 "Strongly Disagree".
  School-level data were analyzed using ED School Climate Surveys (EDSCLS) platform which produces a benchmarked scale score. The benchmarked scale scores were created using item parameters based on a Rasch model. The EDSCLS produced scores which may fall into one of three categories:
  * Least Favorable (scores below 300)
  * Favorable (scores 300-400)
  * Most Favorable (scores above 400-500)
  Additional information on the benchmark scale score calculation is available at safesupportivelearning.ed.gov/edscls/benchmarks
Time Frame: Once annually, spring of each intervention year (2020, 2021, 2022, 2023)
Population: Participants in this outcome measure are schools, because this is a school-level variable. A total of 10 schools participated in each condition. In Spring 2020 and Spring 2021, only one school district participated due to the impact of the novel coronavirus pandemic and related transition to remote learning. In some cases, no teachers or staff responded to the invitation to participate (as indicated in participation numbers below).
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Schools
Arm/Group | Wellness Condition | Partnership
Number analyzed (Participants) | 2590 | 2284
Number analyzed (Schools) | 10 | 10
score on a scale
  Spring 2020 - student: number analyzed (Participants) | 317 | 309
  Spring 2020 - student: number analyzed (Schools) | 5 | 5
  Spring 2020 - student | 289.8 (15.3) | 297.5 (6.8)
  Spring 2020- teacher: number analyzed (Participants) | 80 | 62
  Spring 2020- teacher: number analyzed (Schools) | 8 | 7
  Spring 2020- teacher | 284.2 (30.8) | 270.5 (27.3)
  Spring 2020 - staff: number analyzed (Participants) | 50 | 19
  Spring 2020 - staff: number analyzed (Schools) | 7 | 6
  Spring 2020 - staff | 282.6 (17.6) | 281.0 (18.0)
  Spring 2021 - student: number analyzed (Participants) | 282 | 366
  Spring 2021 - student: number analyzed (Schools) | 5 | 5
  Spring 2021 - student | 267.9 (19.9) | 283.6 (20.9)
  Spring 2021 - teacher: number analyzed (Participants) | 116 | 78
  Spring 2021 - teacher: number analyzed (Schools) | 5 | 5
  Spring 2021 - teacher | 258.8 (31.2) | 250.7 (17.4)
  Spring 2021 - staff: number analyzed (Participants) | 78 | 36
  Spring 2021 - staff: number analyzed (Schools) | 5 | 5
  Spring 2021 - staff | 254.6 (16.6) | 258.8 (9.4)
  Spring 2022 - student: number analyzed (Participants) | 675 | 491
  Spring 2022 - student: number analyzed (Schools) | 10 | 9
  Spring 2022 - student | 289.2 (14.9) | 299.6 (23.6)
  Spring 2022 - teacher: number analyzed (Participants) | 154 | 136
  Spring 2022 - teacher: number analyzed (Schools) | 9 | 9
  Spring 2022 - teacher | 270.4 (19.5) | 278.2 (14.4)
  Spring 2022 - staff: number analyzed (Participants) | 69 | 58
  Spring 2022 - staff: number analyzed (Schools) | 9 | 9
  Spring 2022 - staff | 276.2 (22.9) | 267.9 (26.2)
  Spring 2023 - student: number analyzed (Participants) | 588 | 582
  Spring 2023 - student | 296.3 (22.0) | 305.3 (22.3)
  Spring 2023 - teacher: number analyzed (Participants) | 127 | 84
  Spring 2023 - teacher: number analyzed (Schools) | 9 | 6
  Spring 2023 - teacher | 271.1 (14.4) | 266.2 (15.6)
  Spring 2023 - staff: number analyzed (Participants) | 54 | 63
  Spring 2023 - staff: number analyzed (Schools) | 9 | 7
  Spring 2023 - staff | 269.8 (27.4) | 276.3 (29.3)

4. Primary Outcome: Change in Access to Services
Description: Average number of clinical sessions per student during study enrollment, divided by type (in-person and via tele-health)
Time Frame: Duration of study enrollment from intake to study exit (average 6 months)
Population: Number of students who participated in therapy (attended sessions with provider)
Measure: Mean (Standard Deviation); unit: total number of sessions
Arm/Group | Wellness Condition | Partnership
Number analyzed (Participants) | 578 | 505
total number of sessions
  In-person sessions | 6.12 (7.82) | 6.17 (6.71)
  Telehealth sessions | .83 (2.88) | 1.62 (4.83)

5. Primary Outcome: Change in Client Satisfaction With Services
Description: Client Satisfaction Questionnaire-8 (CSQ-8): 8-item measure for youth 11 and older and adults to assess individual's satisfaction with counseling services. Responses are given using a Likert scales ranging from 1 (indicating poor quality or dissatisfaction with service) to 4 (excellent or highly satisfied with service). Responses were summed for a possible score ranging from 8 to 32; with high scores indicating greater levels of satisfaction for respondents. Analysis included students who completed at least 80% of the items on the scale.
Time Frame: At 3 months and 6 months post-intake
Population: There was some variance in number of students completing measures across the different measures
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wellness Condition | Partnership
Number analyzed (Participants) | 448 | 378
score on a scale
  3 months post intake | 26.90 (3.80) | 27.23 (3.96)
  6 months post intake: number analyzed (Participants) | 378 | 323
  6 months post intake | 27.14 (4.03) | 27.46 (3.97)

6. Primary Outcome: Change in Social Functioning of Students Receiving Services
Description: Child and Adolescent Social and Adaptive Functioning Scale (CASAFS): 24-item measure on school performance, peer relations, family relations, and home duties/self-care. The items range from 0 "Never" to 3 "Always". For some items, "Does not apply to me" is an optional response. Scores were summed for a possible range of 0 to 72, and respondents with at least 80% of items answered were included in analysis. Several items on the instrument required reverse coding prior to analysis. For this scale, lower scores indicate worse outcomes.
Time Frame: Baseline (intake) and at 3 months and 6 months post-intake
Population: There was some variance in number of students completing measures across the different measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wellness Condition | Partnership
Number analyzed (Participants) | 607 | 546
score on a scale
  Intake | 2.05 (0.47) | 2.03 (0.45)
  3 months post intake: number analyzed (Participants) | 452 | 380
  3 months post intake | 2.10 (0.43) | 2.06 (0.45)
  6 months post intake: number analyzed (Participants) | 383 | 324
  6 months post intake | 2.13 (0.47) | 2.08 (0.47)

7. Primary Outcome: Change in Therapeutic Alliance
Description: Therapeutic Alliance Scale for Children-revised (TASC) is a twelve item scale measuring the therapeutic alliance across treatment. The scale is a 12-item, 4-point Likert scale, with responses ranging from 0 "not like me" to 3 "very much like me". Five items on the scale required reverse coding prior to analysis. The total score is the sum of all items, ranging from 0 to 48, where higher scores mean stronger therapeutic alliance (better outcomes). Survey data were collected at 3- and 6-months post intake.
Time Frame: Baseline (intake), and 3 months and 6 months post-intake
Population: There was some variance in number of students completing measures across the different measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wellness Condition | Partnership
Number analyzed (Participants) | 448 | 378
score on a scale
  3 months post intake | 26.90 (3.80) | 27.23 (3.96)
  6 months post intake: number analyzed (Participants) | 378 | 323
  6 months post intake | 27.14 (4.03) | 27.46 (3.97)

8. Primary Outcome: Change in Academic Attendance Rates
Description: School-level variable representing average number of days absent for all students in grades 6-8. The average is calculated by dividing the number of days absent by the total number of days in the school year (180). Note: attendance data are drastically skewed due to the impact of COVID-19. Many schools around the country, including those in one participating district, offered remote-only instruction (no in-person learning) during the 2020-2021 school year; thus the concept of "absence" from school was distorted. Therefore data presented here during 2019-2020 and 2020-2021 may not be meaningfully interpreted.
Time Frame: Annual following each school year (2019-2020, 2020-2021, 2021-2022, and 2022-2023)
Population: Complete attendance records for all students enrolled in grades 6-8 at each of the 20 participating schools
Measure: Mean (Standard Deviation); unit: Absent rate (days absent/days total)
Arm/Group | Wellness Condition | Partnership
Number analyzed (Participants) | 10 | 10
Absent rate (days absent/days total)
  2018-2019 | .083 (.022) | .096 (.056)
  2019-2020 | .051 (.011) | .057 (.025)
  2020-2021 | .345 (.212) | .381 (.237)
  2021-2022 | .162 (.034) | .165 (.056)
  2022-2023 | .122 (.025) | .129 (.037)

9. Secondary Outcome: Change in Mental Health Knowledge
Description: The Guide Curriculum Assessment (GCA): Mental Health Knowledge scale includes 14 true-false questions related to mental health. These items were scored based on the number of correct answers (0 to 14), where higher scores means more correct answers.
Time Frame: Baseline (intake), and 3 months and 6 months post-intake
Population: There was some variance in number of students completing measures across the different measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wellness Condition | Partnership
Number analyzed (Participants) | 603 | 546
score on a scale
  Intake | 5.77 (2.71) | 6.77 (2.74)
  3 months post intake: number analyzed (Participants) | 449 | 385
  3 months post intake | 6.06 (2.78) | 6.74 (3.09)
  6 months post intake: number analyzed (Participants) | 377 | 326
  6 months post intake | 6.02 (2.74) | 6.75 (3.01)

10. Secondary Outcome: Change in Perceived Stigma
Description: The Guide Curriculum Assessment (GCA): Perceived Stigma scale includes 12 items with responses on a 7-point Likert scale from 1 "strongly agree" to 4 "not sure" to 7 "strongly disagree". Two items require reverse coding. Lower scores on this scale mean more stigma and higher scores are optimal, indicating less mental health stigma. Scores on this scale range from 12 (most stigma) to 84 (least stigma).
Time Frame: Baseline (intake), 3 months post intake, and 6 months post intake
Population: There was some variance in number of students completing measures across the different measures
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wellness Condition | Partnership
Number analyzed (Participants) | 604 | 543
score on a scale
  Intake | 65.19 (10.95) | 65.93 (10.58)
  3 months post intake: number analyzed (Participants) | 455 | 381
  3 months post intake | 65.26 (11.42) | 67.52 (10.51)
  6 months post intake: number analyzed (Participants) | 307 | 325
  6 months post intake | 66.68 (10.72) | 68.56 (9.90)

11. Secondary Outcome: Change in Family-school-community Partnerships
Description: Parent Participation Engagement Measure is a 5-item measure of parent participation in therapy sessions, with responses on a 5-point Likert scale ranging from 1 "not at all" to 5 "very much"; and where 0 indicates "not applicable". Scores on this scale can range from 0 to 25 with higher scores indicating higher rates of parent engagement.
Time Frame: At 3 months and 6 months post-intake
Population: There was some variance in number of students completing measures across the different measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wellness Condition | Partnership
Number analyzed (Participants) | 422 | 376
score on a scale
  3 months post intake | 2.44 (1.42) | 2.43 (1.37)
  6 months post intake: number analyzed (Participants) | 366 | 320
  6 months post intake | 2.50 (1.39) | 2.53 (1.39)

ADVERSE EVENTS:
Time Frame: Enrollment into the study (for student self-reported data) was conducted on a rolling basis, beginning in September 2019. Enrollees completed surveys at three intervals: upon intake, three months post-intake, and six months post-intake. After enrollment concluded in June 2023, post-intake assessments were completed through December 2023.
Description: Definitions are as established by Clinical Trials.
Arm/Group | Wellness Condition | Partnership
All-Cause Mortality (participants affected / at risk) | 0/665 | 0/614
Serious Adverse Events (participants affected / at risk) | 0/665 | 0/614
Other Adverse Events (participants affected / at risk) | 0/665 | 0/614

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT03901274/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT03901274/ICF_001.pdf